CLINICAL TRIAL: NCT06108947
Title: Implementing Screening for Preeclampsia in Norway With Aspirin Discontinuation at 24-28 Weeks - a Randomized Controlled Trial
Brief Title: Screening for Preeclampsia in Norway With Aspirin Discontinuation at 24-28 Weeks
Acronym: PEScreenNor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 639348
Record Dates: First submitted 2023-10-17; First posted 2023-10-31 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Active Comparator): Aspirin 150 mg per day from pregnancy week 12 to 36 - according to current recommendations
  Interventions: Drug: Aspirin
- Aspirin discontinuation (Experimental): Discontinuation of Aspirin around 24-28 weeks in low risk women
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin discontinuation
  Other Names: acetyl salicylic acid

SUMMARY:
Study population Around 3500 pregnant women attending a routine ultrasound scan at 11-14 weeks at St. Olavs hospital, Trondheim, Norway.

Study period Dec 2023 - Jul 2025

Screening Patient history, blood pressure, uterine artery mean PI and PlGF will be plotted in the FMF algorithm for screening for preeclampsia in the first trimester. Standardized blood pressure will be measured by trained personnel. Ultrasound scans will be performed by FMF certified doctors and midwives working at the Center for Fetal Medicine in Trondheim. Placenta growth factor (PLGF) will be analyzed with Kryptor technology at Center for Laboratory Medicine, St. Olavs hospital.

Prophylaxis Women with high risk for preterm preeclampsia (risk > 1:100) will be offered aspirin prophylaxis 150 mg x 1 from 11-14 weeks to 36 weeks. Women will be offered to participate in a randomized controlled trial (RCT).

Study design and participants in the RCT A single center, open label, randomized, noninferiority trial conducted at St. Olavs hospital, Trondheim Norway from Dec 2023 to Jul 2025. The investigators will include around 300 women 18 years or older with a singleton live fetus, gestational age between 24 and 28 weeks, high risk of preterm preeclampsia (>1/100) in the first trimester screening, aspirin treatment with a dose 150 mg per day initiated at 16+6 weeks of gestation or less until randomization with a adherence of at least 50% and low SFlt-1/PlGF ratio (Kryptor technology with cut-off 66).

Randomization and masking Between 24 and 28 weeks of gestation, participants will be randomly designed, with a computer-based system in a 1:1 ratio, to continue aspirin (control group) or discontinue aspirin (intervention group). This is an open-label study without masking of patients or providers.

Follow-up Both groups will have visits every 4 weeks between randomization and 36 weeks, and standard antenatal care after 37 weeks until delivery. Treatment adherence will be assessed by patient self-report and tablet count, and fetal growth and Doppler will be assessed at the scheduled visits between randomization and 36 weeks (at 24, 28, 32 and 36 weeks), and according to clinical judgement by obstetricians at the outpatient clinic of the hospital. Women will have a telephone/video link follow-up 1-2 months after birth

DETAILED DESCRIPTION:
The implementation study is divided into four parts/study questions

1. Is screening for preeclampsia cost-effective in a Norwegian setting?

   Folkehelseinstituttet (FHI) in Norway has done a health technology assessment including a cost-effectiveness analysis of introducing screening for preeclampsia at 11-14 weeks in Norway. FHI concluded that 173 cases of preterm preeclampsia could be prevented annually in Norway, and that 17 MNOK could be saved every year. Calculations were based on data from the Norwegian Medical Birth Registry. In this analysis the estimated extra time for measuring the mean uterine artery PI and calculating individual risk was set to 15 min, and costs for analyzing blood samples were set to 600 NOK per woman.

   The present study will assess if the estimated prerequisites in the FHI cost-effectiveness analysis are correct in a clinical setting. The investigators will register time during ultrasound scans and time used for calculating risks and informing patients. Costs for laboratory analyses will be studied. A new cost-effectiveness analysis will be performed if the prerequisites in the previous analysis are far from the ones collected from a clinical setting.
2. Is the blood pressure measured at the general practioner's (GP's) office equivalent to standardized measured BP at the hospital?

   Norwegian women are offered a visit at the GP's office around pregnancy week 8-12. At this visit women are given general information, BP is measured, and blood samples are drawn.

   Most women bring their antenatal chart with information on background, BP and blood samples when the women attend a routine ultrasound scan at 11-14 weeks. The investigators will measure BP at the hospital in a standardized way and compare BPs from the hospital recordings with the antenatal chart. The investigators will study time used for measuring BP in a standardized way at the hospital. If information from the antenatal chart can be used instead of collecting this information again at the hospital visit, the scheduled time can be shortened.
3. Compliance of aspirin use during pregnancy in Norway

   It has been shown that the beneficial effect of aspirin prophylaxis is dependent on compliance. The Aspre trial found a beneficial effect of screening among women using >90% of the prescribed medication.

   The investigators will study compliance among Norwegian women. The investigators estimate that around 300 women will be screen positive and offered aspirin prophylaxis during pregnancy. Women will be asked about aspirin use in pregnancy and tablets will be counted. Women will be stratified according to compliance groups; good (> 90%), intermediate (50-89%) or poor (< 50%) and compared for outcomes of the study.
4. Aspirin discontinuation at 24-28 weeks - a randomized controlled trial

One randomized controlled trial on aspirin discontinuation at 24 to 28 weeks' gestation in pregnancies at high risk of preterm preeclampsia has recently been published. The study included 936 participants and found an incidence of preterm preeclampsia of 1,48% in the intervention group and 1,73% in the control group (absolute difference, -0,25%; 95% CI -1.86% to 1.36) indicating noninferiority to aspirin continuation. The authors stated: "Aspirin treatment should be restricted to pregnant individuals at actual high risk of preeclampsia and administered during the shortest possible time". Furthermore: "given the low incidence of complications of different doses and durations of treatment should be investigated in further studies".

The investigators will do a similar randomized controlled trial. This study will not be sufficiently powered to demonstrate significant differences in preterm preeclampsia between groups (primary outcome), but it may contribute to a pool of similar trials, and can be included in future systematic reviews.

Study design and participants A single center, open label, randomized, noninferiority trial conducted at St. Olavs hospital, Trondheim Norway from Dec 2023 to Jul 2025 will include around 300 women 18 years or older with a singleton live fetus, gestational age between 24 and 28 weeks, high risk of preterm preeclampsia (>1/100) in the first trimester screening, aspirin treatment with a dose 150 mg per day initiated at 16+6 weeks of gestation or less until randomization with a adherence of at least 50% and low SFlt-1/PlGF ratio (Kryptor technology with cut-off 66).

Randomization and masking Between 24 and 28 weeks of gestation, participants will be randomly designed, with a computer-based system in a 1:1 ratio, to continue aspirin (control group) or discontinue aspirin (intervention group). This is an open-label study without masking of patients or providers.

Follow-up Both groups will have visits every 4 weeks between randomization and 36 weeks, and standard antenatal care after 37 weeks until delivery. Treatment adherence will be assessed by patient self-report and tablet count, and fetal growth and Doppler will be assessed at the scheduled visits between randomization and 36 weeks (at 24, 28, 32 and 36 weeks), and according to clinical judgement by obstetricians at the outpatient clinic of the hospital. Women will have a telephone/video link follow-up 1-2 months after birth.

Outcomes Primary outcome is delivery due to preeclampsia before 37 weeks of gestation (preterm preeclampsia).

Secondary outcomes include preeclampsia before 34 weeks of gestation, preeclampsia after 37 weeks of gestation or any other adverse pregnancy outcome, such as severe gestational hypertension, small for gestational age (10th centile or 3rd centile), stillbirth, placental abruption, spontaneous preterm delivery without preeclampsia or gestational hypertension, postpartum hemorrhage, antenatal bleeding, and poor neonatal outcomes.

Ethics A written informed consent will be obtained from all participants. The Regional Committee for Medical and Health Research Ethics in Central Norway (REK-midt) approved the study (REK-midt 639348 and REK - midt 634179).

The study will be registered in Clinicaltrials.gov (639348)

Funding and sponsors The study is funded by Helse-Midt Norge RHF. The funding source has played no role in design of the study and will have no role in data collection, analyses, interpretation or publication.

Participants Kjell Å. B. Salvesen, professor, MD, Phd, Project leader Hanne Mørch, consultant, MD, Phd candidate Ingrid Alsos Lian, consultant, MD, Phd Christian Tappert, consultant, MD

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* singleton live fetus with gestational age between 24 and 28 weeks
* woman with high risk of preterm preeclampsia (>1/100) in the first trimester screening
* aspirin treatment with a dose 150 mg per day initiated at 16+6 weeks of gestation or less until randomization with adherence of at least 50%
* low SFlt-1/PlGF ratio (Kryptor technology with cut-off 66) measured at 24-28 weeks

Exclusion Criteria

* not speaking Norwegian or English language
* fetal anomalies diagnosed with ultrasound
* informed consent for participation in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with preterm preeclampsia | Pregnancy week 24 to pregnancy week 37
  Delivery due to preeclampsia before 37 weeks of gestation

SECONDARY OUTCOMES:
Number of patients with preeclampsia before 34 weeks | Pregnancy week 24 to pregnancy week 34
  Delivery due to preeclampsia before 34 weeks of gestation
Number of patients with preeclampsia after 37 weeks | Pregnancy week 24 to pregnancy week 42
  Delivery with the diagnosis preeclampsia after 37 weeks
Number of patients developing severe gestational hypertension | Pregnancy week 24 to pregnancy week 42
  Delivery with the diagnosis of severe gestational hypertension
Number of patients diagnosed as small for gestational age (10th centile) | Birthweight at delivery between 24 and 42 weeks
  Birthweight defined as SGA below 10th centile
Number of patients diagnosed as small for gestational age (3rd centile) | Birthweight at delivery between 24 and 42 weeks
  Birthweight defined as SGA below 3rd centile
Number of patients diagnosed with placental abruption | Delivery between 24 and 42 weeks
  Diagnosis of placental abruption at delivery- no/yes
Number of patients with spontaneous preterm delivery | Delivery between 24 and 42 weeks
  spontaneous preterm delivery without preeclampsia or gestational hypertension
Number of patients with mild post partum hemorrhage | Delivery between 24 and 42 weeks
  Post partum hemorrhage > 500 ml
Number of patients with severe post partum hemorrhage | Delivery between 24 and 42 weeks
  Post partum hemorrhage > 1000 ml
Number of patients with antenatal bleeding | Pregnancy week 24 to pregnancy week 42
  No/yes
Days of antenatal bleeding | Pregnancy week 24 to pregnancy week 42
  Days of bleeding
Severity of of antenatal bleeding | Pregnancy week 24 to pregnancy week 42
  Maternal hemoglobin measured before delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Å Salvesen, Professor, Principal Investigator — St. Olavs Hospital
Locations (1):
- St. Olavs hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for individual participant data meta-analysis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After completion of the study in Dec 2025
Access Criteria: Contact the principal investigator

REFERENCES:
- [Background] Mendoza M, Bonacina E, Garcia-Manau P, Lopez M, Caamina S, Vives A, Lopez-Quesada E, Ricart M, Maroto A, de Mingo L, Pintado E, Ferrer-Costa R, Martin L, Rodriguez-Zurita A, Garcia E, Pallarols M, Vidal-Sagnier L, Teixidor M, Orizales-Lago C, Perez-Gomez A, Ocana V, Puerto L, Millan P, Alsius M, Diaz S, Maiz N, Carreras E, Suy A. Aspirin Discontinuation at 24 to 28 Weeks' Gestation in Pregnancies at High Risk of Preterm Preeclampsia: A Randomized Clinical Trial. JAMA. 2023 Feb 21;329(7):542-550. doi: 10.1001/jama.2023.0691. PMID 36809321